CLINICAL TRIAL: NCT00154817
Title: A Phase II Clinical and Mechanistic Study of Radiotherapy for Locally Advanced Hepatocellular Carcinoma
Brief Title: A Phase II Study of Radiotherapy for Locally Advanced Hepatocellular Carcinoma (HCC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Health Research Institutes, Taiwan (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 910704
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2005-11-22 (Estimated); Status verified 2002-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: radiotherapy; dynamic contrast enhanced MRI; hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiotherapy

INTERVENTIONS:
Procedure: radiotherapy

SUMMARY:
1. This is a phase II study of radiotherapy for patients with locally advanced HCC.
2. Patients whose tumor(s) are not suitable for other local treatment, such as surgery, trans-arterial chemoembolization (TAE), ethanol injection, or radiofrequency ablation. will be enrolled.
3. Radical radiotherapy will be started after pre-treatment evaluation. The total dose of RT will be 50Gy in 25 fractions to local tumor(s).
4. Dynamic contrast enhanced MRI and serum samples will be done at the following time points to assess the change in tumor perfusion: (1) before the start of thalidomide treatment; (2) 2weeks after radiotherapy begins; and (3) 1 month after radiotherapy completes. DCEMRI will then be done every 3 months until disease progression.
5. The study was designed to evaluate the response rate and tolerability of radical radiotherapy for locally advanced HCC. The sample size was determined by the expected incidence of grade 4 toxicity and response rate of radiotherapy for locally advanced HCC. Since the grade 4 toxicity of radiotherapy alone is 10%, the response rate is 60% we need at least 12 patients to evaluate for the treatment.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is one of the most common malignancies in Asian countries. Surgical resection is potentially the only form of curative treatment. However, less than 20% of patients are surgical candidates at diagnosis. Nonsurgical treatment options include transcatheter arterial chemoembolization (TACE), percutaneous acetic acid or ethanol injection therapy and radio-frequency ablation. They are sometimes unsatisfactory, especially for patients with portal vein thrombosis or large infiltrative hepatic tumors. Repeated treatments are often necessary.

Radiotherapy (RT) for the treatment of HCC has been attempted for more than 4 decades. Early trials adopted whole liver irradiation but used an inadequate radiation dose. Because of the unsatisfactory results obtained with this low-dose whole liver irradiation, RT has not long been considered for the treatment of HCC. Recently, local, not whole, liver RT has been attempted by several investigators, who have shown that high doses of radiation can be safely delivered to a portion of the liver alone or in combination with other nonsurgical modalities. Their results suggest that local RT can be an effective component of the treatment regimen for HCC.

Development of surrogate markers to monitor the response of HCC to radiotherapy is important because of the following reasons. First, the response as evaluated by conventional imaging studies is usually slow and may be unreliable. The maximal response to radiotherapy is often achieved 6 months after completion of radiotherapy. The slow response to radiotherapy makes it difficult to modify an ineffective treatment regimen in a more timely fashion to HCC, especially for patients with low serum a-fetal protein (AFP). Second, intra-hepatic recurrence outside RT field is a common cause of RT treatment failure. Nearly half of the patients recur after RT with lesions outside RT fields. Inflammation and normal liver damage caused by RT may have deleterious effect on tumor control through the release of cytokines or angiogenic factors. Therefore, the biological consequence of RT in both the tumors and the non-tumor liver parenchyma shall be carefully evaluated.

Dynamic contrast enhanced magnetic resonance imaging (DCEMRI) may assess hepatic perfusion parameters which correlate with the severity of cirrhosis and portal hypertension. In cervical cancer, DCEMRI enables us to evaluate the microcirculation of tumors as well as the blood perfusion of normal parenchyma. Malignancy, stage and prognosis have all been correlated with the enhancement parameters in cervical, breast cancers.Several studies have shown that successful therapies also result in changes in DCEMRI parameters, which may prove to be a more accurate and earlier indication of response. De Vries et al reported, in rectal carcinoma patients receiving preoperative radiotherapy, that perfusion index showed a significant increase in the 1st and 2nd week of treatment. High perfusion index values correlated with greater lymph node down-staging. Moffat et al also reported increased apparent diffusion coefficient (ADC) 3 weeks after the initiation of RT in brain cancer patients who had better local response. Circulating angiogenic factors have been shown to provide important prognostic information about a variety of cancers (21). Elevated serum levels of VEGF or bFGF have been associated with increased invasiveness of HCC. Placental growth factor (PlGF), a homolog of VEGF, has been shown to have a synergistic effect with VEGF in pathologic angiogenesis, such as angiogenesis induced by cancer or ischemia, but its prognostic value in human cancers remains unclear.

We would like to correlate functional image studies of blood flow and serum cytokines during radiotherapy with treatment outcome in hepatocellular carcinoma patients.

ELIGIBILITY:
Inclusion Criteria:

* 1.1 Patients with measurable, locally advanced HCC that are not suitable for other local therapies, including surgery, TAE, alcohol injection, or radiofrequency ablation.

1.2 Patients with histological confirmed HCC or patients who do not have histological diagnosis but have met all of the following criteria: 1.2.1 Presence of chronic viral hepatitis and/or cirrhosis 1.2.2 Presence of hepatic tumor(s) with image findings (sonography, CT scan) compatible with HCC.

1.2.3 A persistent elevation of serum a-fetoprotein level ³ 400 ng/ml without any evidence of ana-fetoprotein-secreting germ cell tumor.

1.3 Patients without any local or systemic therapy for HCC within 4 weeks. 1.4 Patients with age > 20 years and < 70 years. 1.5 Patients with a performance status of ECOG score < 1. 1.6 Patients must fulfill all of the following criteria: 1.6.1 Child-Pugh's Score ≦ 7. 1.6.2 Serum total bilirubin < 1.5 times upper normal limit (UNL). 1.6.3 Serum alanine transaminase (ALT) < 5 times UNL 1.6.4 Platelet count > 5.0 x 104 / mm3. 1.6.5 White blood cell count > 3,000 / mm3. 1.6.6 Serum creatinine < 2.0 mg/dL 1.7 Patient must have local tumors less than one half of the whole liver and the tumors can be encompassed within RT fields 1.8 Signed informed consent 1.9 Sexually active patients, in conjunction with their partner, must practice birth control during, and for 2 months after, thalidomide therapy.

1.10 Female patients in child-bearing age must have negative pregnancy test.

Exclusion Criteria:2.1. Patients with documented extrahepatic metastasis. 2.2. Patients who received previous radiotherapy to abdominal area. 2.3. Patients who have received thalidomide treatment prior to enrollment. 2.4. Patients who had other investigational drug treatment within 4 weeks prior to enrollment.

2.5. Patients with NCI grade 2 or greater peripheral neuropathy of any causes. 2.6. Patients with other systemic diseases that required concurrent usage of glucocorticosteroid or immunosuppressant agent(s).

2.7. Patients who have major systemic diseases that the attending physicians consider inappropriate for radiotherapy or thalidomide therapy.

-

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12
Dates: Start 2002-01; Study Completion 2005-05

PRIMARY OUTCOMES:
The primary objective is to evaluate response rate, tolerability and failure pattern of local radiotherapy for the treatment of locally advanced HCC.

SECONDARY OUTCOMES:
The second objective is to correlate parameters of tumor perfusion assessed by dynamic contrast enhanced MRI (DCEMRI) and serum cytokine levels with clinical outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Ju Ch'ang, M.D., Principal Investigator — National Health Research Institutes, Division of Cancer Research